CLINICAL TRIAL: NCT06982560
Title: Assessment and Management of Acute Heart Failure Patients Guided by Electrical Cardiometry
Brief Title: Electrical Cardiometry in Management of Acute Heart Failure
Acronym: EC/AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0107959
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Heart Failure (AHF)
Keywords: cardiometry, acute heart failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: traditional group (Placebo Comparator): traditional methods like clinical examination, lung ultrasound, inferior vena cava
  Interventions: Other: traditonal methods
- Group B: cardiometry group (Experimental): use of cardiometry parameters like cardiac output, thoracic fluid content and systemic vascular resistance
  Interventions: Device: electrical cardiometry

INTERVENTIONS:
Device: electrical cardiometry — use of cardiometry parameters as cardiac output, thoracic fluid content, systemic vascular resistance
  Arms: Group B: cardiometry group
Other: traditonal methods — clinical examination, lung ultrasound, inferior vena cava
  Arms: Group A: traditional group

SUMMARY:
The goal of this clinical trial is to assess if electrical cardiometry (EC) could help in managing acute heart failure (AHF). The main questions it aims to answer are:

1. Is there effect of use of cardiometry on rate of use of vasopressors, vasodilators and inotropes?
2. is there effect of use of cardiometry on mortality and hospital length of stay?

Researchers compared cardiometry to traditional methods like clinical examination, lung ultrasound and inferior vena cava.

Participants were divided into two groups, one managed by cardiometry and the other by traditional methods, then followed till improvement or death and compared regarding use of medications, length of stay and mortality

DETAILED DESCRIPTION:
The purpose of the research is to assess the role of electrical cardiometry in hemodynamic monitoring in studied cases with acute heart failure to guide treatment.

This is a prospective controlled research that involved fifty patients, diagnosed with acute heart failure and admitted to critical care units at Alexandria University Hospitals, patients were divided into 2 groups:

Group A: was assessed by traditional methods which include: clinical examination including chest auscultation and systolic blood pressure measurement, lung ultrasound and inferior vena cava assessment and managed according to the results of these parameters.

Group B: was assessed by electrical cardiometry parameters as cardiac output, thoracic fluid content (TFC) and systemic vascular resistance (SVR) and was managed as following: inotropes up and down titration according to cardiac output readings, use of vasopressors or vasodilators according to SVR readings, doses of diuretics were modified according to TFC readings.

ELIGIBILITY:
Inclusion Criteria:

* acute heart failure

Exclusion Criteria:

* pregnant females, atrial fibrillation, severe valvular diseases, skin lesions in thoracic area, large pleural effusion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
mortality and intensive care unit (ICU) length of stay | 7 days
  number of days in ICU and mortality in ICU

SECONDARY OUTCOMES:
use of vasopressors, vasodilators, inotropes | 7 days
  number of patients who needed these medications

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed R Elsalamouny, MD, Principal Investigator — Lecturer of Critical Care Medicine, Alexandria University
Locations (1):
- Alexandria University Hospitals, Alexandria, Alexandria Governorate, Egypt

REFERENCES:
- [Background] Shaheen, Mostafa Mohamed, Ahmed Said Elgebaly, Ghada Fouad Elbaradey, and Amira Mahfouz Alqablawi. 2022. "Fluid Management Using Cardiometry in ARDS Patients". Journal of Advances in Medicine and Medical Research 34 (11):21-27. https://doi.org/10.9734/jammr/2022/v34i1131360.
- [Background] Paranjape VV, Henao-Guerrero N, Menciotti G, Saksena S, Agostinho M. Agreement between Electrical Cardiometry and Pulmonary Artery Thermodilution for Measuring Cardiac Output in Isoflurane-Anesthetized Dogs. Animals (Basel). 2023 Apr 21;13(8):1420. doi: 10.3390/ani13081420. PMID 37106987
- [Background] Abdou , Noura, Heba Elmahdy, Osama Tolba, Nihal Shihab, Asmaa Elmesiry, and Mohammed Rowisha. 2023. "Electrical Cardiometry Versus Echocardiography in Assessment of Hemodynamic Status in Preterm Neonates With Septic Shock". Journal of Advances in Medicine and Medical Research 35 (20):144-55. https://doi.org/10.9734/jammr/2023/v35i205184.
- [Background] Liu YH, Dhakal BP, Keesakul C, Kacmarek RM, Lewis GD, Jiang Y. Continuous non-invasive cardiac output monitoring during exercise: validation of electrical cardiometry with Fick and thermodilution methods. Br J Anaesth. 2016 Jul;117(1):129-31. doi: 10.1093/bja/aew156. No abstract available. PMID 27317712
- See also: Information about cardiometry — https://www.osypkamed.com/technology/noninvasive-hemodynamics/electrical-cardiometry/